CLINICAL TRIAL: NCT06948942
Title: Comparison of Exercise Capacity, Muscle Oxygenation and Physical Activity Levels Between Patients With Interstitial Lung Disease and Healthy Individuals
Brief Title: Exercise Capacity, Muscle Oxygenation, and Physical Activity Between Patients With Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: 2024 - 1689
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Lung Diseases (ILD); Healthy Individuals; Exercise Capacity; Muscle Oxygenation; Physical Activity Level
Keywords: Interstitial lung diseases; Healthy individuals; Exercise capacity; Muscle oxygenation; Physical activity level
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ILD: That group consists of patients who had been diagnosed with ILD by doctors. Oxygen consumption using CPET, muscle oxygenation with a near-infrared spectroscopy device, physical activity level using multi-sensor activity monitor, pulmonary function using spirometer, lower extremity functional exercise capacity with 6MWT, upper-extremity functional exercise capacity with 6PBRT, respiratory muscle strength using mouth pressure device, peripheral muscle strength with hand-held dynamometer, inspiratory muscle endurance using incremental threshold loading test, dyspnea with 'Modified Medical Research Council' Dyspnea Scale and 'Turkish version of London Chest Daily Living Activity Scale', dyspnea at rest, during, and after exercise training with 'Modified Borg Scale', disease-related quality of life with 'Turkish version of Saint George Respiratory Questionnaire' and sleep quality with 'Pittsburg Sleep Quality Index' will be evaluated in patients with ILD.
- Healthy Controls: That group consists of people who have not been diagnosed with a disease. Oxygen consumption using CPET, muscle oxygenation with a near-infrared spectroscopy device, physical activity level using multi-sensor activity monitor, pulmonary function using spirometer, lower extremity functional exercise capacity with 6MWT, upper-extremity functional exercise capacity with 6PBRT, respiratory muscle strength using mouth pressure device, peripheral muscle strength with hand-held dynamometer, inspiratory muscle endurance using incremental threshold loading test, dyspnea with 'Modified Medical Research Council' Dyspnea Scale and 'Turkish version of London Chest Daily Living Activity Scale', dyspnea at rest, during, and after exercise training with 'Modified Borg Scale', disease-related quality of life with 'Turkish version of Saint George Respiratory Questionnaire' and sleep quality with 'Pittsburg Sleep Quality Index' will be evaluated in healthy controls.

SUMMARY:
Interstitial lung diseases (ILD) are a group of chronic respiratory diseases that cause significant mortality and morbidity worldwide. Although there are studies in the literature comparing different lung disease groups with healthy individuals, it has been determined that there is no study comparing the exercise capacity, muscle oxygenation, physical activity level, respiratory functions, respiratory and peripheral muscle strength, inspiratory muscle endurance, quality of life and sleep quality of individuals diagnosed with ILD with healthy individuals.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) are a group of chronic respiratory diseases that cause significant mortality and morbidity worldwide. Patients with interstitial lung disease experience a decrease in both static and dynamic lung volumes and carbon monoxide diffusion capacity (DLCO). As a result of this pathological mechanism, exertional dyspnea and exercise intolerance increase. Therefore, individuals with ILD tend to avoid activities that will increase shortness of breath, which leads to physical inactivity and an increasingly sedentary lifestyle. Due to this vicious cycle, individuals whose functional exercise capacity is also limited become more dependent in daily life activities. In addition, peripheral muscle dysfunction is another important factor that causes exercise intolerance in individuals with all chronic lung diseases, including ILD. Although there are studies in the literature comparing different lung disease groups with healthy individuals, it has been determined that there is no study comparing the exercise capacity, muscle oxygenation, physical activity level, respiratory functions, respiratory and peripheral muscle strength, and inspiratory muscle endurance of individuals with ILD with healthy individuals. The primary aim of our study was to compare the exercise capacity, muscle oxygenation and physical activity levels of patients with interstitial lung disease and healthy individuals. The secondary aim of our study was to compare the respiratory functions, respiratory and peripheral muscle strength, inspiratory muscle endurance, dyspnea, quality of life and sleep quality of patients with interstitial lung disease and healthy individuals.

ELIGIBILITY:
Patients who will participate in the study;

Inclusion Criteria:

* Patients diagnosed with ILD according to ATS/ERS criteria,
* Ages between 18 and 75,
* Pulmonary infection during the previous month,
* Participants who voluntarily participated in the study were included.

Exclusion Criteria:

* Patients were excluded if they had:
* Acute pulmonary exacerbation or respiratory infection in the last four weeks
* Obstructive lung disease
* Systemic conditions affecting neurological, neuromuscular, orthopedic, or physical functions
* Recent participation in a planned exercise program (within three months)
* Cognitive impairment affecting exercise test understanding
* Contraindications to exercise testing per the American Sports Medicine Association
* Cancer, renal, or hepatic disease
* Aortic stenosis, complex arrhythmia, or aortic aneurysm
* Serious cardiovascular diseases like uncontrolled hypertension, diabetes, heart failure, or arrhythmia

For healthy individuals who will participate in the study;

Inclusion Criteria:

* No diagnosed chronic disease,
* Healthy adults between the ages of 45-80

Exclusion Criteria:

* Individuals with a Mini Mental State Assessment Scale score of less than 24,
* A smoking history of at least 10 packs×years or more,
* Having had COVID-19,
* A BMI of >30 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and Male
Study Population: Patients diagnosed with ILDs and healthy individuals
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | Trough study completion, an average of 1 year
  Maximal exercise capacity will be assessed by symptom-limited cardiopulmonary exercise testing on a treadmill at gradually increasing workload, and oxygen consumption will be measured during the test.
Muscle Oxygenation | Trough study completion, an average of 1 year
  Muscle oxygenation before, during and after exercise tests will be measured with a near-infrared spectroscopy device.
Physical Activity Level | Trough study completion, an average of 1 year
  Individuals' physical activity level will be assessed with a multi-sensor physical activity monitor.

SECONDARY OUTCOMES:
Upper extremity functional exercise capacity | Trough study completion, an average of 1 year
  To evaluate upper extremity functional exercise capacity, 6-minute pegboard and ring tests will be applied twice with 15-30 minute intervals. Before the test, individuals will be seated and rested for at least 10 minutes. Individuals will be provided with detailed information about the application of the test before the test. Patients will be informed not to interfere with rings that fall during the test and to continue the test. It will be explained that they can stop and rest if they feel too uncomfortable to continue the test, but this time will be included in the test duration. Before the actual test, subjects will be allowed to move up and down one loop as a practice to learn the test procedure. As a test result, the total number of rings worn at the end of six minutes will be recorded in numbers.
Lower extremity functional exercise capacity | Trough study completion, an average of 1 year
  A 6-minute walking test will be applied according to ATS/ERS criteria to evaluate lower extremity functional exercise capacity.
Dyspnea | Trough study completion, an average of 1 year
  The assessment of dyspnea at rest, during, and after exercise training will be made with the Modified Borg scale. The Modified Borg scale is a subjective scale and scores the shortness of breath at rest and/or during activity between 0-10. The lowest score of 0 (zero) indicates 'none', and the highest score of 10 (ten) indicates 'maximal' shortness of breath. The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living. The London Chest Activities of Daily Living Scale, developed by Garrod et al. to examine dyspnea that occurs with daily living activities in chronic obstructive pulmonary disease and whose Turkish validity and reliability were performed by Saka et al., will be used to assess shortness of breath that occurs during activities of daily living.
Respiratory Muscle Strength | Trough study completion, an average of 1 year
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Inspiratory muscle endurance | Trough study completion, an average of 1 year
  The increasing threshold load using the inspiratory muscle training device will be evaluated with the respiratory muscle endurance test. The test will be started with 30% of MIP and the inspiratory threshold load will be increased by 10% of MIP every two minutes. The test will be terminated in the presence of severe dyspnea/fatigue or when patients cannot take three deep breaths in a row. At the end of the test, the respiratory muscle endurance result will be obtained by multiplying the maximal inspiratory pressure (cmH2O) that the patients can maintain for one minute and the total time (seconds).
Peripheral muscle strength | Trough study completion, an average of 1 year
  Shoulder abductor and knee extansor muscle strength will be assessed with a portable handheld dynamometer (JTECH Power Track Commander, Baltimore, USA).
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (Forced vital capacity (FVC)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (FEV1/FVC) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.
Disease Related Quality of life | Trough study completion, an average of 1 year
  The Saint George Respiratory Questionnaire is a questionnaire used to assess the quality of life in respiratory diseases and its Turkish validity and reliability were conducted by Polatlı et al. The questionnaire consists of 3 sections: symptoms (8 items), activities (16 items), and effects of the disease (26 items) and a total of 50 items: The 3 sections of the test are scored separately. Then, a total score is obtained. The total score varies between 0-100. A score of zero is normal, while a score of 100 indicates maximum disability. As the total score increases, it indicates that the patients' quality of life is poor.
Sleep quality | Trough study completion, an average of 1 year
  The Pittsburgh Sleep Quality Index will be used to evaluate the patients' sleep quality. It contains a total of 24 questions. 19 of these questions are answered by the individual by evaluating himself/herself. The remaining 5 questions are answered by the individual's bed partner or roommate, if any. The questionnaire includes questions asked under 7 main headings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping pills and daytime functions. Each of these 7 main headings is first evaluated within itself. Then, the scores of the 7 components are added. If the total score is over 5 points, it is considered as poor sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Nazire Nur YILDIZ, M.Sc., Principal Investigator — Nigde Omer Halisdemir University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Principal Investigator — Gazi University; Beyzanur ÖYMEZ, Principal Investigator — Gazi University; Ayşenur GÜVENİR, M.Sc., Principal Investigator — Yozgat Bozok University; Nilgün YILMAZ DEMİRCİ, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To protect patient data, it will not be shared.

REFERENCES:
- See also: Ward J, McDonald C. Interstitial lung disease - An approach to diagnosis and management. Aust Fam Physician. 2010;39(3):106-10. PubMed PMID: 20369109. — https://pubmed.ncbi.nlm.nih.gov/20369109/
- See also: Cakmak A, Inal-Ince D, Sonbahar-Ulu H, Bozdemir-Ozel C, Ozalp O, Calik-Kutukcu E, et al. Physical activity of patients with bronchiectasis compared with healthy counterparts: A cross-sectional study. Heart Lung. 2020;49(1):99-104. Epub 20190914. doi: 10. — https://pubmed.ncbi.nlm.nih.gov/31530430/
- See also: Arikan H, Yatar I, Calik-Kutukcu E, Aribas Z, Saglam M, Vardar-Yagli N, et al. A comparison of respiratory and peripheral muscle strength, functional exercise capacity, activities of daily living and physical fitness in patients with cystic fibrosis and — https://pubmed.ncbi.nlm.nih.gov/26241869/
- See also: Fırat M, Mutlu Ş, Yoleri B, Boşnak Güçlü M. Comparison of respiratory functions, muscle strength, and physical activity among children with primary ciliary dyskinesia with and without Kartagener's syndrome and healthy controls. Physiother Theory Pract. 2 — https://pubmed.ncbi.nlm.nih.gov/38018157/
- See also: Garcia T, Mantoani LC, Silva H, Zamboti CL, Ribeiro M, Ramos EMC, et al. Characteristics of Skeletal Muscle Strength in Subjects With Interstitial Lung Disease. Arch Phys Med Rehabil. 2024;105(6):1099-105. Epub 20240124. doi: 10.1016/j.apmr.2024.01.006. — https://pubmed.ncbi.nlm.nih.gov/38272247/
- See also: Wallaert B, Monge E, Le Rouzic O, Wémeau-Stervinou L, Salleron J, Grosbois J-M. Physical activity in daily life of patients with fibrotic idiopathic interstitial pneumonia. Chest. 2013;144(5):1652-8. — https://pubmed.ncbi.nlm.nih.gov/23928896/